CLINICAL TRIAL: NCT03705494
Title: A Feasibility Randomised Controlled Study of an Innovative Postnatal Breastfeeding Peer Counselling Programme
Brief Title: Home-based Breastfeeding Peer Counselling Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BFPC1
Record Dates: First submitted 2018-09-02; First posted 2018-10-15 (Actual); Results first posted 2020-12-24 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2019-09

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Peer counsellor
MeSH Terms: conditions — Breast Feeding | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based peer counselling intervention (Active Comparator): Women planning to breastfeed who meet the study's inclusion criteria
  Interventions: Other: Home-based peer counselling (web-based) intervention
- Standard usual care (No Intervention): Women planning to breastfeed who meet the study's inclusion criteria

INTERVENTIONS:
Other: Home-based peer counselling (web-based) intervention — The intervention consists of 5-6 home based visits (web-based) over 6 months by trained peer counsellors who will focus on breastfeeding among mothers who have already decided to breastfeed and are interested in this programme.
  Arms: Home-based peer counselling intervention

SUMMARY:
A feasibility study is proposed in the current study as women who had given birth to their first babies recruited to a previous project specifically expressed the need for postnatal breastfeeding support from peer counsellors at home and there is evidence that this could be of benefit for women and their infants. Evidence of whether women in Hong Kong who had peer counsellors have better breastfeeding outcomes compared to women who had standard care however is not available. Prior to undertaking a definitive trial, the investigators need to know if women would be willing to be recruited and randomised to an intervention or standard care.

DETAILED DESCRIPTION:
Peer counselling and support has been shown to be effective in improving breastfeeding (BF) initiation, duration and exclusiveness. Peer counselling is being introduced into different country settings worldwide as an intervention to support women to achieve successful commencement and maintenance of breastfeeding, given the range of health benefits for the woman and her infant. Findings from one Cochrane review suggested that postnatal contacts in the home may reduce infant health service utilisation in the weeks following the birth, and that more home visits may encourage more women to exclusively breastfeed.

The planned study A feasibility randomized controlled trial (RCT) study is proposed in the current study as women who had given birth to their first babies recruited to a previous project specifically expressed the need for postnatal BF support from peer counsellors at home and there is evidence that this could be of benefit for women and their infants. Evidence of whether women in Hong Kong who had peer counsellors have better breastfeeding outcomes compared to women who had standard care however is not available. Prior to undertaking a definitive RCT, the investigators need to know if women would be willing to be recruited and randomised to an intervention or standard care.

This study is important for several reasons. Chinese women are expected to be housebound during the first month postnatally due to the tradition of 'doing the month', when problems with infant feeding and/or infants failing to thrive due to poor feeding could result in a decision to stop breastfeeding. The innovative home-based intervention the investigators will undertake will address an important service gap in Hong Kong to promote and sustain exclusive breastfeeding, and could be an effective strategy which reflects Chinese culture. The Health Care and Promotion Scheme grant review panel recommended that although an evaluation of a home-based peer counselling project is a high priority, a small-scale feasibility study was needed before a definitive RCT application is submitted.

Peer counsellors will be recruited from those who passed the UNICEF and La Leche League Peer Counselling Training programme. Additional training tailored to issues that they may encounter in home-based contacts with women who are breastfeeding, for example solving problems of exclusive breastfeeding and correct breastfeeding technique will be needed and conducted by team leaders for the peer counsellors. Women planning to breastfeed who meet the study's inclusion criteria will be recruited from hospital postnatal ward and randomly allocated using opaque, sealed envelopes, by an independent research assistant not involved in participant recruitment, data collection or analysis to the intervention group (n=10, home-based peer counselling intervention and standard usual care) and control groups (n=10, standard usual care).

ELIGIBILITY:
Inclusion Criteria:

* Primiparous mothers
* Intention to breastfeed
* Singleton pregnancy
* Term infant (37-42 weeks gestational)
* Cantonese speaking
* Hong Kong resident
* Mother with no serious medical or obstetrical complications.

Exclusion Criteria:

* infant is <37 weeks gestation,
* infant has an Apgar score <8 at five minutes,
* infant has a birthweight <2500 grams,
* infant has any severe medical conditions or congenital malformations
* infant is placed in the special care baby unit for more than 48 hours after birth
* infant is placed in the neonatal intensive care unit at any time after birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kris YW Dr Lok, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lok KY, Chow CLY, Shing JSY, Smith R, Lam CCO, Bick D, Chang YS. Feasibility, acceptability, and potential efficacy of an innovative postnatal home-based breastfeeding peer support programme in Hong Kong: a feasibility and pilot randomised controlled trial. Int Breastfeed J. 2021 Apr 13;16(1):34. doi: 10.1186/s13006-021-00381-5. PMID 33849582

RESULTS

PARTICIPANT FLOW:
Groups:
- Home-based Peer Counselling Intervention: Women planning to breastfeed who meet the study's inclusion criteria
  Home-based peer counselling intervention: The intervention consists of 5-6 home based visits over 6 months by trained peer counsellors who will focus on breastfeeding among mothers who have already decided to breastfeed and are interested in this programme.
Period: Overall Study
Arm/Group | Home-based Peer Counselling Intervention | Standard Usual Care
Started | 10 | 10
Completed | 3 | 7
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home-based Peer Counselling Intervention | Standard Usual Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Count of Participants; unit: Participants]
  18-24 years | 3 | 0 | 3
  25-29 years | 1 | 1 | 2
  30-34 years | 4 | 6 | 10
  ≥35 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 10 | 10 | 20
Maternal education [Count of Participants; unit: Participants]
  Primary | 0 | 0 | 0
  Compulsory Secondary | 0 | 1 | 1
  Post-secondary | 5 | 4 | 9
  University Degree | 4 | 5 | 9
  Post-graduate Degree | 1 | 0 | 1
Monthly family income [Count of Participants; unit: Participants]
  <HK$15,000 | 1 | 1 | 2
  HK$15,000-29,999 | 2 | 1 | 3
  ≥HK$30,000 | 7 | 8 | 15
Length of residence in Hong Kong [Count of Participants; unit: Participants]
  <5 years | 0 | 1 | 1
  5-15 years | 0 | 0 | 0
  ≥15 years | 10 | 9 | 19
Return to work postpartum [Count of Participants; unit: Participants]
  No or not sure | 3 | 1 | 4
  Yes | 7 | 9 | 16
Parity [Count of Participants; unit: Participants]
  Primiparous | 9 | 8 | 17
  Multiparous | 1 | 2 | 3
Self-breastfed [Count of Participants; unit: Participants] | 4 | 6 | 10
Attended antenatal childbirth class [Count of Participants; unit: Participants] | 8 | 8 | 16
Attended antenatal breastfeeding class [Count of Participants; unit: Participants] | 7 | 7 | 14
Planned to exclusively breastfeed [Count of Participants; unit: Participants] | 9 | 8 | 17
Planned duration of breastfeeding [Count of Participants; unit: Participants]
  <6 months | 1 | 0 | 1
  ≥6 months | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing Qualitative Interviews on the Peer Counselling Breastfeeding Intervention
Description: The number of participants who have completed the in-depth qualitative interviews on their views on the peer counselling breastfeeding intervention programme.
  Participants who are in the intervention group and have received intervention were approached for qualitative interviews after study completion at six months. Eight participants have received intervention, two of which has been lost to follow-up. Thus, six participants were approached for the interview. One participants refused to be interviewed.
Time Frame: through study completion, an average of 6 months
Population: Participants in the intervention group who have received peer support intervention or completed the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Peer Counselling Intervention | Standard Usual Care
Number analyzed (Participants) | 6 | 0
Participants
  Completed qualitative interview | 5 | 0
  Not completed qualitative interview | 1 | 0

2. Secondary Outcome: Number of Participants Who Exclusively Breastfeed
Description: The number of participants who exclusive breastfeed at each follow-up time-points
Time Frame: At 1, 2, 4 and 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Peer Counselling Intervention | Standard Usual Care
Number analyzed (Participants) | 10 | 10
Participants
  1 month postpartum | 4 | 3
  2 months postpartum | 3 | 3
  4 months postpartum | 3 | 3
  6 months postpartum | 1 | 1

3. Secondary Outcome: Exclusive Breastfeeding Duration
Description: Exclusive breastfeeding duration is measured using time in weeks
Time Frame: At 1, 2, 4 and 6 months postpartum
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Home-based Peer Counselling Intervention | Standard Usual Care
Number analyzed (Participants) | 10 | 10
weeks | 6.0 (9.1) | 4.7 (8.0)

4. Secondary Outcome: Women's Self-efficacy in Breastfeeding
Description: Breastfeeding Self-efficacy Scale measures maternal breastfeeding self-efficacy. It consists of 14 items measured on a 5-point likert scale. On scale 1 indicates "not at all confident" and 5 indicates "always confident". Total scores range from 14 to 70 with higher scores indicating greater breastfeeding confidence and self-efficacy.
Time Frame: At baseline, 2 and 4 months postpartum
Population: Cases lost to follow-up or withdrew were not included in the follow-up assessments. Cases who were no longer breastfeeding at the time of follow-up were not also not included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Peer Counselling Intervention | Standard Usual Care
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 37.1 (10.8) | 44.5 (5.9)
  2 months postpartum: number analyzed (Participants) | 7 | 8
  2 months postpartum | 45.3 (12.7) | 46.6 (13.2)
  4 months postpartum: number analyzed (Participants) | 4 | 6
  4 months postpartum | 47.3 (11.8) | 57.5 (13.7)

5. Secondary Outcome: Women's Attitude in Breastfeeding
Description: Iowa Infant Feeding Attitude Scale is a measure of attitudes towards feeding. It consists of 17 items that are scored on a 5-point Likert scale, which ranges from 1 (strongly disagree) to 5 (strongly agree). Eight items are worded in a favourable manner towards breastfeeding, while nine are favourable towards formula feeding. Items favouring formula feeding are reverse-scored (i.e. 1=5, 2=4, 4=2 and 5=1). The total attitude scores range from 17 (indicating positive bottle feeding attitudes) to 85 (reflecting positive breastfeeding attitudes). Total scores are grouped into the following three categories: (1) positive towards breastfeeding (70-85); (2) neutral (49-69); and (3) positive towards formula feeding (17-48).
Time Frame: At baseline, 2 and 4 months postpartum
Population: Cases lost to follow up or withdraw are not included
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Peer Counselling Intervention | Standard Usual Care
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 66.2 (6.2) | 61.5 (5.2)
  2 months postpartum: number analyzed (Participants) | 9 | 8
  2 months postpartum | 59.3 (7.3) | 63.1 (8.4)
  4 months postpartum: number analyzed (Participants) | 8 | 8
  4 months postpartum | 61.5 (6.0) | 66 (7.3)

ADVERSE EVENTS:
Time Frame: 6 months or between participants' recruitment and exit the study.
Arm/Group | Home-based Peer Counselling Intervention | Standard Usual Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03705494/Prot_SAP_000.pdf